CLINICAL TRIAL: NCT05118399
Title: Addition of Liposomal Bupivacaine to Standard Bupivacaine Versus Standard Bupivacaine Alone in the Supraclavicular Brachial Plexus Block: a Randomized Controlled Trial
Brief Title: Analgesic Effect of Liposomal Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW21-046
Record Dates: First submitted 2021-11-01; First posted 2021-11-12 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- To receive supraclavicular BPB using standard ropivacaine only. (Active Comparator): 20ml of plain bupivacaine will be injected using 2 syringes, so 10ml of 0.5% plain bupivacaine will be injected, and immediately followed by another 10ml of 0.5% plain bupivacaine.
  Interventions: Drug: Bupivacaine Injection [Marcaine]
- To receive supraclavicular BPB using liposomal bupivacaine together with ropivacaine. (Experimental): 10ml of 0.5% plain bupivacaine will be injected, and immediately followed by 10ml of 1.33% liposomal bupivacaine.
  Interventions: Drug: Bupivacaine Liposome 13.3 MG/ML [Exparel]

INTERVENTIONS:
Drug: Bupivacaine Injection [Marcaine] — Bupivacaine injection [Marcaine] is the standard treatment used in our hospital.
  Arms: To receive supraclavicular BPB using standard ropivacaine only.
Drug: Bupivacaine Liposome 13.3 MG/ML [Exparel] — Bupivacaine liposome is a multivesicular formulation of bupivacaine that allows rapid absorption and prolonged release of bupivacaine.
  Arms: To receive supraclavicular BPB using liposomal bupivacaine together with ropivacaine.

SUMMARY:
Brachial plexus blocks (BPB) are commonly used to provide regional anaesthesia for patients undergoing distal radial fracture surgery. Distal radial (DR) fracture surgery is a commonly performed orthopaedic surgery, and is usually associated with moderate postoperative pain. Poor postoperative pain control can impair rehabilitation, delay recovery and negatively impact outcomes after surgery. Liposomal bupivacaine (EXPAREL) is a multivesicular formulation of bupivacaine that allows rapid absorption and prolonged release of bupivacaine. Liposomal bupivacaine can provide longer analgesia for up to 72 hours, and may therefore achieve greater analgesic efficacy compared to non-liposomal long-acting local anaesthetics. A number of clinical trials have studied the effect liposomal bupivacaine given as local infiltration. However, there is little evidence on liposomal bupivacaine for regional nerve blocks, and the use of liposomal bupivacaine for supraclavicular brachial plexus block - which is used for regional anaesthesia for distal radial fracture surgery - have not been studied before. This project is a randomized controlled trial to determine whether adding liposomal bupivacaine to long-acting local anaesthetics for supraclavicular BPB will improve and prolong postoperative analgesia in patients undergoing distal radial fracture surgery. Longer term secondary outcomes would be accessed including upper limb functional scores, chronic pain, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) status I-III
* Age 18-90 years old
* Scheduled for distal radial fracture fixation (Open reduction and internal fixation with volar approaching locking plate)
* Patients with informed consent to participate in the study

Exclusion Criteria:

* Ulnar shaft/ neck physis fracture
* Revision surgery
* Previous fractures or surgery in the affected distal radius
* Surgery involving more than the affected arm
* Higher energy and high-grade fracture cases - road traffic accident, fall from height, open fractures, combined distal radius and distal ulna fractures, fractures requiring external fixation, fractures with severe articular comminution or severe metaphyseal extension, comminuted fractures requiring more than a single volar approach incision and a single volar locking plate implant
* Cases with painful conditions affecting the upper limb prior to surgery such as cervical spine, shoulder, elbow, other hand and wrist problems
* Cases with baseline (pre-injury) QuickDASH score worse than 10 out of 100
* Respiratory compromise (requires long term oxygen)
* History of seizures
* Pre-existing neurological disorder/deficit
* Chronic opioid user (use for 3 months or more)
* Presence of chronic pain condition (pain duration over 3 months)
* Alcohol or substance abuse
* Psychiatric illness
* Impaired mental state
* Local infection
* Allergy to analgesic drugs: local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs), opioids
* Impaired renal function (defined as effective glomerular filtration rate less than 30ml/min/1.73m2
* Impaired liver function (defined as plasma bilirubin over 34micromol/L; international normalized ratio [INR] 》／=1.7, alanine aminotransferase [ALT] over 100U/L, aspartate aminotransferase [AST] over 100U/L)
* Coagulopathy (platelet count 《100,000/ml and/or INR 》／=1.5) or the use of anticoagulants (not including aspirin) that precludes the use of supraclavicular BPB
* Pregnancy
* Patient refusal for regional nerve blocks
* Patient refusal to join the clinical trial
* Patient unable/unwilling to attend post-op rehabilitation programme
* Injury on duty

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
postoperative AUC pain score at rest | First 48 hours after surgery
  Pain severity would be rated at rest after surgery using numerical rating scale with 0 to 10 where 0=no pain and 10=the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong